CLINICAL TRIAL: NCT00374777
Title: FK199B (Zolpidem MR Tablet) Phase III Clinical Study -A Double-Blind, Placebo- and Nitrazepam-Controlled, Group-Comparison Study in Patients With Insomnia Associated With Schizophrenia and Manic-Depressive Psychosis
Brief Title: A Double-blind, Group-comparison P-III Study With Zolpidem MR Using Placebo and Nitrazepam in Insomnia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6199-CL-0008
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Insomnia; schizophrenia; manic-depressive psychosis; zolpidem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Schizophrenia; Bipolar Disorder | interventions — Nitrazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: zolpidem MR
- 2 (Experimental)
  Interventions: Drug: zolpidem MR
- 3 (Active Comparator)
  Interventions: Drug: nitrazepam
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zolpidem MR — oral
  Other Names: FK199B
  Arms: 1; 2
Drug: nitrazepam — oral
  Arms: 3
Drug: placebo — oral
  Arms: 4

SUMMARY:
A multicenter, randomized, double-blind, triple-dummy, group-comparison study using placebo and nitrazepam as a comparative drug.

ELIGIBILITY:
Inclusion Criteria:

* Nonorganic insomnia associated with schizophrenia and manic-depressive psychosis.

Exclusion Criteria:

* Patients with allergic reactions to zolpidem or nitrazepam; Patients with serious cardiac disorders; serious hepatic impairment; serious renal diseases.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean wake time after sleep onset during the double-blind period | 2 Weeks

SECONDARY OUTCOMES:
Mean total sleep time during the double-blind period | 2 Weeks
Mean number of nightly awakenings during the double-blind period | 2 Weeks
Mean sleep latency during the double-blind period | 2 Weeks
Patient impression during the double-blind period | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- Japan (6):
  - Chubu Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region